CLINICAL TRIAL: NCT04145050
Title: Carbohydrate Oxidation in Elite Wheelchair Racers During Marathon Simulation
Acronym: COW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Nicholas Burd, Primary Investigator, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20020
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Dietary Carbohydrate; Para-Athletes

STUDY DESIGN:
Intervention Model Description: Randomized, Cross-Over
Who Masked: Participant, Investigator
Masking Description: Participants as well as researchers will not be informed of trial intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carbohydrate Dose: 0 grams carbohydrate (Experimental): Participants will be randomly selected, in a cross-over fashion, to ingest 0 grams/hour, 30 grams/ hour, or 60 grams/ hour of carbohydrate beverage throughout each experimental trial.
  Interventions: Other: Carbohydrate dosing
- Carbohydrate Dose: 30 grams carbohydrate (Experimental): Participants will be randomly selected, in a cross-over fashion, to ingest 0 grams/hour, 30 grams/ hour, or 60 grams/ hour of carbohydrate beverage throughout each experimental trial.
  Interventions: Other: Carbohydrate dosing
- Carbohydrate Dose: 60 grams carbohydrate (Experimental): Participants will be randomly selected, in a cross-over fashion, to ingest 0 grams/hour, 30 grams/ hour, or 60 grams/ hour of carbohydrate beverage throughout each experimental trial.
  Interventions: Other: Carbohydrate dosing

INTERVENTIONS:
Other: Carbohydrate dosing — The purpose of this study is to examine effects of different carbohydrate doses during marathon simulation in elite wheelchair racers.

SUMMARY:
To examine the effect of varying amounts of carbohydrate ingestion on performance, gastrointestinal experiences, and other physiological markers in elite wheelchair racers during a simulated marathon.

DETAILED DESCRIPTION:
The metabolic demands created by endurance activities, which include muscle and liver glycogen depletion as well as losses in body fluids and electrolytes, are significant limitations to the performance potential of the athlete. For this reason, a well-supported recommendation exists for such athletes to consume a carbohydrate (CHO) formula, in particular, one containing electrolytes during their activity. Furthermore, the current CHO recommendations to support prolonged activity have been developed specifically for able-bodied athletes, thus are potentially inappropriate for para athletes.

Metabolic and physiological functions are altered in individuals with physical disabilities, so it is unknown how transferable these recommendations are to para athletes. As such, it is important to understand this population's unique carbohydrate requirements for performance optimization.

Recently, our group showed stable elevated circulating glucose concentrations by utilizing two different sources of CHO dosed at 60 g/h when compared to water. Significantly improved performance was observed with both CHO conditions. These findings, combined with studies showing decreased net muscle glycogen degradation during intravenous glucose infusion (3.5 g/min), show the importance of plasma glucose concentration for sustained performance. Therefore, the purpose of this study is to investigate the SCI-specific responses to exogenous CHO during a full marathon simulation (MS).

Twelve highly trained men and women (20-50 yrs old) will be recruited to the study. The inclusion criteria are: 1.) Best marathon time lower than 2h 2.) and ≥6 months of prior training history. After initial screenings, participants will perform three marathon (MS) trials. In cross-over trials, each subject will participate in a MS trial consisting of a challenge (90% of subject's best marathon time) followed by a time trial (TT) representing the last 10% of the marathon time. During each MS trial, participants will be randomly assigned to receive either water, 30g, or 60g of carbohydrate (CHO) every 15 minutes in the form of a sports nutrition beverage. Repeated blood and breath sampling will occur throughout the MS. These samples will be used to determine glucose concentration, lactate concentration, as well as CHO and fat oxidation. Heart rate, core temperature, blood pressure, ratings of perceived exertion and GI symptoms will also be assessed throughout the MS and after the time trial.

Completion of this research study will help to identify more appropriate CHO recommendations for para athletes to support prolonged endurance exercise. This will aid in the understanding of the unique physiological and metabolic needs of para athletes as compared to their able-bodied counterparts, thus enhancing inclusivity within sports nutrition literature.

ELIGIBILITY:
Inclusion Criteria:

* < 2-hour best marathon time

  * 6 months prior training history

Exclusion Criteria:

* - Chronic Smoking or tobacco use
* Active cardiovascular disease
* Diabetes Mellitus or other metabolic disorders
* Liver kidney, or urinary disease
* Musculoskeletal/Orthopedic disorders (e.g., osteoarthritis, rheumatoid arthritis, tendinitis, gout, fibromyalgia, patellar tendinopathy, or chronic low back pain)
* Neuromuscular disorders
* hypertension
* Diagnosed GI tract diseases
* Heart Disease
* Neurological disease
* Epilepsy
* Respiratory disease
* Pregnancy
* Contraindications for exercise
* <6 months of prior training history

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Performance | 10-15 minutes
  Performance will be measured by time required to complete a 2.6 mile time-trial immediately following marathon simulation

SECONDARY OUTCOMES:
Ratings of gastrointestinal (GI) experiences | Throughout experimental protocol for 1.5 - 2 hours
  Using a visual analog scale (Visual Analog Symptom Scale), participants will record GI symptoms (from 0-100 whereby higher numbers indicate worse experiences) at various time points throughout experimental trial
Blood Glucose Concentration | Throughout experimental protocol for 1.5 - 2 hours
  Blood glucose concentration will be measured at various time points throughout experimental trial
Blood Lactate Concentration | Throughout experimental protocol for 1.5 - 2 hours
  Blood lactate concentration will be measured at various time points throughout experimental trials
Core Temperature | Throughout experimental protocol for 1.5 - 2 hours
  Core temperature will be measured at various time points throughout experimental trials via ingestible thermometer sensors
Rated Perceived Exertion (RPE) | Throughout experimental protocol for 1.5 - 2 hours
  RPE, or how hard an athlete feels they are working, will be recorded at various time points throughout the experimental trial

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Burd, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Disability Rehababilitation and Education Services, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Data will be coded and de-identified.